CLINICAL TRIAL: NCT03744728
Title: Randomized Trial of Fast Bacterial Identification and Phenotypic Antimicrobial Susceptibility Testing in Patients With Positive Blood Cultures Using the Accelerate PhenoTest™ BC Kit, Performed on the Accelerate Pheno™ System as Compared With the Verigene® BC-GP/GN
Brief Title: Genotypic Versus Phenotypic Susceptibility Testing of Positive Blood Cultures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Accelerate Diagnostics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ECP000001
Record Dates: First submitted 2018-11-15; First posted 2018-11-16 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Bloodstream Infection
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Accelerate Pheno (Active Comparator): Fast ID and AST of positive blood culture bottles using the Accelerate PhenoTest™ BC kit with the Accelerate Pheno™ System
  Interventions: Diagnostic Test: Accelerate PhenoTest™ BC kit
- Standard of Care (Active Comparator): Standard culture and AST of positive blood culture bottles plus the Verigene® BC-GP/GN
  Interventions: Diagnostic Test: Standard of Care

INTERVENTIONS:
Diagnostic Test: Accelerate PhenoTest™ BC kit — The Accelerate PhenoTest™ BC kit with the Accelerate Pheno™ System is a fully-integrated in vitro diagnostic system. It is FDA-cleared to perform ID of bacteria and yeast in less than 90 minutes and AST in less than 7 hours, on average, directly from positive blood culture
  Arms: Accelerate Pheno
Diagnostic Test: Standard of Care — Standard culture and AST of positive blood culture bottles plus the Verigene® BC-GP/GN
  Other Names: Verigene® BC-GP/GN
  Arms: Standard of Care

SUMMARY:
This study is designed as a prospective, randomized, open-label trial evaluating antimicrobial utilization, clinical outcomes, and healthcare costs among patients with positive blood cultures. Patients will be randomized to one of the following FDA-cleared devices that will be used to assess the workflow impact of fast identification (ID) and antimicrobial susceptibility testing (AST) in the microbiology lab and in the quality of care in patients: 1) Standard culture and AST of positive blood culture bottles plus the Verigene® Blood Culture Gram-positive/Gram-negative kit (BC-GP/GN); or 2) Fast ID and AST of positive blood culture bottles using the Accelerate PhenoTest™ BC kit with the Accelerate Pheno™ System.

ELIGIBILITY:
Inclusion Criteria:

* All positive blood cultures (including on-panel/off-panel/contaminants) identified during local laboratory business hours
* All adult (≥18 years of age)

Exclusion Criteria:

* Identification of blood culture positivity outside of local laboratory business hours (e.g. whenever laboratories are staffed to perform both rapid testing and routine testing)
* Positive blood culture in the prior week with same Gram stain result
* Transferred from an outside hospital and had a history of a previously positive blood culture of the same Gram stain result
* Previously enrolled in the study
* Only the first positive culture for each patient will be included during the study period; any subsequent episode of bloodstream infection (BSI) will be excluded
* Died or were transitioned to comfort care within 24 hours of enrollment
* Negative Gram-stain
* Not admitted to hospital for ≥ 24 hours following blood culture positivity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 774 (Actual)
Dates: Start 2019-05-23 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Duration of anti-pseudomonal β-lactam therapy | 4 days after randomization
  Mean duration of anti-pseudomonal β-lactam therapy
Duration of anti-methicillin-resistant Staphylococcus aureus (MRSA) therapy | 4 days after randomization
  Mean duration of MRSA therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Hennepin County Medical Center, Minneapolis, Minnesota, United States